CLINICAL TRIAL: NCT03008252
Title: Lactose Intolerance and Cow's Milk Protein Allergy in Non-celiac Wheat Sensitivity Patients
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Pasquale Mansueto, MD, University of Palermo
Other Study IDs: ACPM12
Record Dates: First submitted 2016-12-29; First posted 2017-01-02 (Estimated); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Non-celiac Wheat Sensitivity
Keywords: Non-celiac wheat sensitivity; lactose intolerance; cow's milk protein allergy
MeSH Terms: conditions — Lactose Intolerance; Milk Hypersensitivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Lactose breath test — Lactose breath test in NCWS patients with symptoms related to milk and/or milk derivates ingestion.
Other: DBPC cow's milk protein challenge — DBPC cow's milk protein challenge in NCWS patients with symptoms related to milk and/or milk derivates ingestion.

SUMMARY:
In the last few years a new clinical entity has emerged which includes patients who consider themselves to be suffering from problems caused by wheat and/or gluten ingestion, even though they do not have celiac disease (CD) or wheat allergy. This clinical condition has been named non-celiac gluten sensitivity (NCGS), although in a recent article, the researchers suggested the term "non-celiac wheat sensitivity" (NCWS), because it is not known to date what component of wheat actually causes the symptoms. The clinical picture of NCWS is characterized by combined gastrointestinal (bloating, abdominal pain, diarrhea and/or constipation, nausea, epigastric pain, gastroesophageal reflux, aphthous stomatitis) and extra-intestinal or systemic manifestations (headache, depression, anxiety, 'foggy mind,' tiredness, dermatitis or skin rash, fibromyalgia-like joint/muscle pain, leg or arm numbness, and anemia). Lactose intolerance and cow's milk protein allergy (CMPA) are two medical conditions with a very high prevalence in the general population, and there is a large overlap between NCWS symptoms and lactose intolerance and CMPA symptoms. Therefore, the aims of the present study are to investigate 1) the prevalence of positive lactose breath test and DBPC cow's milk protein challenge in NCWS patients with self-reported gastrointestinal symptoms related to milk and/or milk derivates ingestion, 2) the clinical, serological, and histological characteristics of NCWS patients with lactose intolerance and CMPA in comparison to NCWS patients without lactose intolerance and CMPA.

DETAILED DESCRIPTION:
In the last few years, a new clinical entity has emerged which includes patients who consider themselves to be suffering from problems caused by wheat and/or gluten ingestion, even though they do not have celiac disease (CD) or wheat allergy. This clinical condition has been named non-celiac gluten sensitivity (NCGS), although in a recent article, the researchers suggested the term "non-celiac wheat sensitivity" (NCWS), because it is not known to date what component of wheat actually causes the symptoms. Other areas of doubt in NCWS regard its pathogenesis, while some papers reported intestinal immunologic activation, others linked NCWS to the dietary short chain carbohydrate (fermentable oligo-di-monosaccharides and polyols, FODMAPs) load. The researchers recently demonstrated that higher proportions of patients with NCWS develop autoimmune disorders, are antinuclear antibodies (ANA) positive, and show DQ2/DQ8 haplotypes compared with patients with irritable bowel syndrome (IBS), supporting an immunologic involvement in NCWS. The clinical picture of NCWS is characterized by combined gastrointestinal (bloating, abdominal pain, diarrhea and/or constipation, nausea, epigastric pain, gastroesophageal reflux, aphthous stomatitis) and extra-intestinal or systemic manifestations (headache, depression, anxiety, 'foggy mind,' tiredness, dermatitis or skin rash, fibromyalgia-like joint/muscle pain, leg or arm numbness, and anemia). Lactose intolerance and cow's milk protein allergy (CMPA) are two conditions with a very high prevalence in the general population and there is a large overlap between NCWS and lactose intolerance and CMPA symptoms. Therefore, the aims of the present study are to investigate 1) the prevalence of positive lactose breath test and DBPC cow's milk protein challenge in NCWS patients with self-reported gastrointestinal and extra-intestinal symptoms related to milk and/or milk derivates ingestion, 2) the clinical, serological, and histological characteristics of NCWS patients with lactose intolerance and CMPA in comparison to NCWS patients without lactose intolerance and CMPA.

ELIGIBILITY:
Inclusion Criteria:

All the NCWS patients will meet the recently proposed criteria:

* negative serum anti-tissue transglutaminase and antiendomysium (EmA) IgA and IgG antibodies
* absence of intestinal villous atrophy
* IgE-mediated immunoallergy tests negative to wheat and cow's milk protein (skin prick tests and/or serum specific IgE detection).

Adjunctive criteria adopted in our patients will be:

* resolution of the gastrointestinal and extra-intestinal symptoms on a standard elimination diet, without wheat, cow's milk, egg, tomato, chocolate, or other food(s) causing self-reported symptoms
* symptom reappearance on double-blind placebo-controlled (DBPC) wheat challenge, performed as described previously.

Exclusion Criteria:

Exclusion criteria will be:

* age <18 years
* positive EmA in the culture medium of the duodenal biopsies, even if the villi to crypts ratio in the duodenal mucosa was normal
* self-exclusion of wheat from the diet and refusal to reintroduce it before entering the study
* other organic cutaneous and/or gastrointestinal diseases
* concomitant treatment with steroids and/or antihistamines.

Lactose intolerance and CMPA will be diagnosed, in patients with self-reported gastrointestinal and extra-intestinal symptoms related to milk and/or milk derivates ingestion, using lactose breath test and DBPC cow's milk protein challenge, respectively.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The researchers prospectively will survey adult patients with functional gastroenterological symptoms (Rome III criteria) and a definitive diagnosis of NCWS, referred at the Department of Internal Medicine at the University Hospital of Palermo, Italy, and at the Department of Internal Medicine of the Hospital of Sciacca, Agrigento, Italy, between January 2017 and January 2019, comparing the characteristics of the ones suffering from lactose intolerance and CMPA with those who do not suffer from lactose intolerance and CMPA.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Positive lactose breath test and DBPC cow's milk protein challenge in NCWS patients self-reporting symptoms related to milk and/or milk derivates ingestion. | January 2017 to December 2017
  Prevalence of positive lactose breath test and DBPC cow's milk protein challenge in NCWS patients with self-reported gastrointestinal and extra-intestinal symptoms related to milk and/or milk derivates ingestion.

SECONDARY OUTCOMES:
Lactose intolerance and CMPA in NCWS patients | January 2017 to December 2017
  Frequency of lactose intolerance and CMPA in NCWS patients

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Carroccio, PhD, Study Director — University of Palermo
Locations (2):
- Italy (2):
  - Internal Medicine Department of the Hospital of Sciacca (Agrigento), Sciacca, Agrigento
  - Internal Medicine Department of the University Hospital of Palermo, Palermo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Carroccio A, Mansueto P, Iacono G, Soresi M, D'Alcamo A, Cavataio F, Brusca I, Florena AM, Ambrosiano G, Seidita A, Pirrone G, Rini GB. Non-celiac wheat sensitivity diagnosed by double-blind placebo-controlled challenge: exploring a new clinical entity. Am J Gastroenterol. 2012 Dec;107(12):1898-906; quiz 1907. doi: 10.1038/ajg.2012.236. Epub 2012 Jul 24. PMID 22825366
- [Result] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Non-celiac gluten sensitivity: literature review. J Am Coll Nutr. 2014;33(1):39-54. doi: 10.1080/07315724.2014.869996. PMID 24533607
- [Result] Carroccio A, Rini G, Mansueto P. Non-celiac wheat sensitivity is a more appropriate label than non-celiac gluten sensitivity. Gastroenterology. 2014 Jan;146(1):320-1. doi: 10.1053/j.gastro.2013.08.061. Epub 2013 Nov 22. No abstract available. PMID 24275240
- [Result] Carroccio A, D'Alcamo A, Mansueto P. Nonceliac wheat sensitivity in the context of multiple food hypersensitivity: new data from confocal endomicroscopy. Gastroenterology. 2015 Mar;148(3):666-7. doi: 10.1053/j.gastro.2014.11.047. Epub 2015 Jan 24. No abstract available. PMID 25625764
- [Result] Carroccio A, Soresi M, D'Alcamo A, Sciume C, Iacono G, Geraci G, Brusca I, Seidita A, Adragna F, Carta M, Mansueto P. Risk of low bone mineral density and low body mass index in patients with non-celiac wheat-sensitivity: a prospective observation study. BMC Med. 2014 Nov 28;12:230. doi: 10.1186/s12916-014-0230-2. PMID 25430806
- [Result] Mansueto P, Seidita A, D'Alcamo A, Carroccio A. Role of FODMAPs in Patients With Irritable Bowel Syndrome. Nutr Clin Pract. 2015 Oct;30(5):665-82. doi: 10.1177/0884533615569886. Epub 2015 Feb 18. PMID 25694210
- [Result] Carroccio A, Brusca I, Mansueto P, D'alcamo A, Barrale M, Soresi M, Seidita A, La Chiusa SM, Iacono G, Sprini D. A comparison between two different in vitro basophil activation tests for gluten- and cow's milk protein sensitivity in irritable bowel syndrome (IBS)-like patients. Clin Chem Lab Med. 2013 Jun;51(6):1257-63. doi: 10.1515/cclm-2012-0609. PMID 23183757
- [Result] Carroccio A, Montalto G, Custro N, Notarbartolo A, Cavataio F, D'Amico D, Alabrese D, Iacono G. Evidence of very delayed clinical reactions to cow's milk in cow's milk-intolerant patients. Allergy. 2000 Jun;55(6):574-9. doi: 10.1034/j.1398-9995.2000.00417.x. PMID 10858991
- [Result] Carroccio A, Montalto G, Cavera G, Notarbatolo A. Lactose intolerance and self-reported milk intolerance: relationship with lactose maldigestion and nutrient intake. Lactase Deficiency Study Group. J Am Coll Nutr. 1998 Dec;17(6):631-6. doi: 10.1080/07315724.1998.10718813. PMID 9853544